CLINICAL TRIAL: NCT03797287
Title: Arthroscopic Transosseous vs. Anchored Rotator Cuff Repair: A Randomized Clinical Trial
Brief Title: Arthroscopic Transosseous vs. Anchored Rotator Cuff Repair
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: IRB will be terminated
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: IRB00046834
Record Dates: First submitted 2019-01-07; First posted 2019-01-09 (Actual); Last update posted 2019-05-30 (Actual); Status verified 2019-05

CONDITIONS: Shoulder Pain Chronic; Shoulder Pain; Rotator Cuff Tear; Rotator Cuff Injury
MeSH Terms: conditions — Shoulder Pain; Rotator Cuff Injuries

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Tensor Tunnler (Experimental): The Tensor Tunneler (Chattanooga, TN) will be used to create the bone tunnels during the arthroscopic procedure. This is an FDA approved device and is used currently in routine clinical practice.
  Interventions: Device: Tensor Tunnler
- Smith and Nephew PEEK Helicoil Anchor (Active Comparator): The anchors used in this trial are FDA approved and are used currently in routine clinical practice (Anchor Rotator Cuff Repair).
  Interventions: Procedure: Anchor Rotator Cuff Repair

INTERVENTIONS:
Device: Tensor Tunnler — Create the bone tunnels during the arthroscopic rotator cuff repair procedure
  Arms: Tensor Tunnler
Procedure: Anchor Rotator Cuff Repair — The suture anchors (Smith and Nephew PEEK Helicoil Anchor) are inserted in bone and the sutures are then used to sew the tendons to bone arthroscopically.
  Arms: Smith and Nephew PEEK Helicoil Anchor

SUMMARY:
This study will compare arthroscopic transosseous versus anchored rotator cuff repairs in terms of clinical outcomes, rotator cuff integrity, and cost-effectiveness. With the collection of patient-reported outcomes the health of patients undergoing each rotator cuff repair technique will be assessed. The aims of this study will be achieved through a clinical randomized controlled trial and a cost-effectiveness analysis.

DETAILED DESCRIPTION:
Study Design: After the decision to proceed with arthroscopic rotator cuff repair, patients will be asked to participate in this prospective randomized clinical trial.

Study Procedures:

Before Surgery: The Informed Consent process will be completed prior to any data collection. Consent will be completed after explanation of each treatment group and the data to be collected. Baseline and demographic data will be collected prior to surgery:

Randomization: Subjects will be randomized prior to surgery into one of the two rotator cuff repair technique groups using REDCap software. Randomization will be stratified by gender.

Patient Visits:

Patients will complete their questionnaires and testing before surgery then within 2 weeks, 3 months, 6 months, 1 year, and 2 years After the first week of surgery, patients will be given a pain diary to record all narcotic pain medications they consume during the 1st week post-op.

An ultrasound will be done during their 6 month, 1 year, and 2 year follow up.

ELIGIBILITY:
Inclusion Criteria:

* Adults age 18-75 years old
* Full thickness rotator cuff tears of any size (documented by MRI or ultrasound)
* Patients planning surgical repair with Dr. Uma Srikumaran (PI of this study) at Johns Hopkins Shoulder Service (Columbia, Odenton Clinic sites; Howard County General Hospital/Bayview/Johns Hopkins Hospital operative sites)

Exclusion Criteria:

* Patients with partial tears, massive rotator cuff tears that are irreparable, isolated subscapularis tears, and associated pathology (advanced degenerative changes)
* Patients undergoing revision rotator cuff tears will be excluded.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-02-01 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Change in condition of the shoulder as assessed by American Shoulder and Elbow Surgeon (ASES) Score | Before surgery, 2 weeks, 3 months, 6 months, and 1 year after surgery
  10 separate questions is scored on an ordinal scale from 0-3 for a maximal raw functional score of 30 (no difficulties).

SECONDARY OUTCOMES:
Change in shoulder pain as assessed by Visual Analog Pain Score | Before surgery, 2 weeks, 3 months, 6 months, and 1 year after surgery
  Patients are asked to identify whether they are having pain in the shoulder and are asked to record the location of their pain on a 10 cm line that ranges from 0(no pain at all) to 10 (pain as bad as it can be)
Change in Range of Motion (ROM) | Before surgery, within 1 month after surgery, 3 months, 6 months, 1 year
  Total (combined glenohumeral and scapulothoracic) shoulder motion is measured. Both active and passive motion for both shoulders is recorded. Forward elevation is measured as the maximum arm-trunk angle viewed from any direction. External rotation is measured with the arm comfortably at the side and also with the arm at 90° of abduction. Internal rotation is measured by noting the highest segment of spinal anatomy reached with the thumb. Cross-body adduction is measured by measuring the distance of the antecubital fossa from the opposite acromion.
Change in Strength Testing | Before surgery, 2 weeks, 3 months, 6 months, and 1 year after surgery
  Strength is graded according to the Medical Research Council grade. Strength is measured in forward elevation, abduction, external rotation with the arm comfortably at the side, and internal rotation with the arm comfortably at the side. A perfect score is a 5 in each category.
Change in quality of life as assessed by the Western Ontario Rotator Cuff (WORC) Index | Before surgery, 1 year after surgery, 2 years after surgery
  Quality of Life Measurement tool for patients with rotator cuff disease where patients mark a line on 21 visual analogue scale (VAS) lines labeled 0 (not affected) - 100 (affected). These items will ask about physical symptoms, sports and recreation, work, social function, and emotions. The maximum score is 2100 for worst possible symptoms and 0 represents no symptoms at all.
Change in health related quality of life as assessed by Short-Form Six-Dimension (SF-6D) | Before surgery, 2 weeks, 3 months, 6 months, and 1 year after surgery
  Measures of health related quality of life (HRQoL) using 11 items from the SF-36 or SF-12. Patients are asked about their physical functioning, role limitations, social functioning, pain, mental health, and vitality. A score of 1 represents full health.
Implant Cost | Within 1 month after surgery
  Review of costs through our billing department

CONTACTS AND LOCATIONS:
Overall Officials: Uma Srikumaran, MD, MBA, Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins, Columbia, Maryland, United States

IPD SHARING:
Plan to Share IPD: Undecided